CLINICAL TRIAL: NCT05112809
Title: Noninvasive Cochlear Stimulation System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Gaurav N. Pradhan, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-007158
Record Dates: First submitted 2021-10-28; First posted 2021-11-09 (Actual); Results first posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: Normal hearing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Normal hearing subjects (Experimental): Subjects with normal hearing will have a standard hearing test utilizing the cochlear stimulation system.
  Interventions: Device: Cochlear Stimulation System (CSS)
- Bilateral hearing impaired (Experimental): Subjects with bilateral hearing impairment will have a standard hearing test utilizing the cochlear stimulation system.
  Interventions: Device: Cochlear Stimulation System (CSS)
- Asymmetrical hearing-impaired (Experimental): Subjects with asymmetrical hearing-impairment will have a standard hearing test utilizing the cochlear stimulation system.
  Interventions: Device: Cochlear Stimulation System (CSS)

INTERVENTIONS:
Device: Cochlear Stimulation System (CSS) — Cochlear stimulation with surround sound and noise cancellation

SUMMARY:
The purpose of this research is to develop a portable wearable hardware headset using a computer-based software that can establish the optimal stimulation parameters appropriate for medical and consumer environments for individuals with hearing impaired and normal hearing individuals.

ELIGIBILITY:
Inclusion Criteria:

- Employee of Mayo Clinic.

Exclusion Criteria:

* Pregnant.
* Cochlear implants.
* History of fluctuating sensorineural hearing loss.
* Skin diseases of the head.
* History of acute paroxysmal tachycardia.
* History of trigeminal neuralgia.
* Recent of paralysis of the facial nerve.
* Recent cerebrovascular stroke.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Cevette, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- [Derived] Kingsbury SE, Cevette MJ, Stepanek J, Pradhan GN. Investigating Speech Intelligibility Capabilities of Electrical Auditory Stimulation. Mil Med. 2025 Sep 3:usaf430. doi: 10.1093/milmed/usaf430. Online ahead of print. PMID 40899906
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal Hearing Subjects | Bilateral Hearing Impaired | Asymmetrical Hearing-impaired
Started | 55 | 5 | 8
Completed | 55 | 5 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Hearing Subjects | Bilateral Hearing Impaired | Asymmetrical Hearing-impaired | Total
Number analyzed (Participants) | 55 | 5 | 8 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.78 (9.33) | 56.8 (11.39) | 59 (13.44) | 38.51 (13.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 3 | 3 | 37
  Male | 24 | 2 | 5 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 2 | 2 | 15
  Not Hispanic or Latino | 37 | 2 | 5 | 44
  Unknown or Not Reported | 7 | 1 | 1 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 0 | 4
  White | 38 | 3 | 8 | 49
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 8 | 1 | 0 | 9
Region of Enrollment [Number; unit: participants]
  United States | 55 | 5 | 8 | 68

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Electric Current Subjects Indicated They Could Hear a Tone at Certain Frequencies
Description: Evaluated by increasing the amplitude of the current input until the subject could hear a tone at 250 Hz, 500 Hz, 1,000 Hz, 2,000 Hz, 4,000 Hz, 8,000 Hz, 10,000 Hz, 12,500 Hz and 16,000 Hz. The mean electric current is reported in Milliampere (mA).
Time Frame: Baseline, approximately 2 hours
Measure: Mean (Standard Deviation); unit: mA
Groups:
- Normal Hearing Subjects: Subjects with normal hearing had a standard hearing test utilizing the cochlear stimulation system.
  Cochlear Stimulation System (CSS): Cochlear stimulation with surround sound and noise cancellation
- Bilateral Hearing Impaired: Subjects with bilateral hearing impairment had a standard hearing test utilizing the cochlear stimulation system.
  Cochlear Stimulation System (CSS): Cochlear stimulation with surround sound and noise cancellation
- Asymmetrical Hearing-impaired: Subjects with asymmetrical hearing-impairment had a standard hearing test utilizing the cochlear stimulation system.
  Cochlear Stimulation System (CSS): Cochlear stimulation with surround sound and noise cancellation
Arm/Group | Normal Hearing Subjects | Bilateral Hearing Impaired | Asymmetrical Hearing-impaired
Number analyzed (Participants) | 55 | 5 | 8
mA
  250 Hz | 2.16 (1.07) | 2.88 (1.44) | 2.88 (0.97)
  500 Hz | 1.86 (1.62) | 2.93 (1.42) | 2.40 (1.14)
  1,000 Hz | 1.09 (0.42) | 1.75 (0.53) | 1.70 (0.42)
  2,000 Hz | 1.29 (0.43) | 1.77 (0.81) | 1.71 (0.60)
  4,000 Hz | 1.56 (0.67) | 3.50 (2.35) | 1.84 (0.68)
  8,000 Hz | 1.71 (0.79) | 2.25 (1.06) | 3.00 (1.76)
  10,000 Hz | 1.97 (1.06) | 3.25 (1.06) | 3.96 (2.51)
  12,500 Hz | 2.29 (1.32) | 6.00 (3.46) | 3.67 (1.47)
  16,000 Hz | 2.94 (1.30) | 5.00 (0.00) | 4.21 (1.25)

2. Primary Outcome: Speech Intelligibility in Quiet Environment
Description: Measured using the modified rhyme test (MRT) consisting of a set of 50 six-item wordlist. Each word list contains single syllable words with a consonant-vowel-consonant sound sequence. Subjects completed electrical word recognition testing in a quiet environment. Electrodes were placed at 3 unique locations (forehead, mastoid, neck) to measure how well speech could be delivered to the subject through the skin electrodes in a manner that would allow subjects to recognize words in a quiet environment. There were 2 experiments done for speech intelligibility. The first involved 20 subjects (outcome 2) and aimed to assess speech intelligibility performance in a basic, quiet environment without background noise. This phase focused on evaluating the fundamental hearing performance. Once it was established that speech intelligibility was satisfactory with electrical stimulation, we proceeded to test an additional 30 subjects in both quiet and noisy environments (outcome 3).
Time Frame: Baseline, approximately 2 hours
Population: MRT was not collected from bilateral hearing impaired and asymmetrical hearing-impaired participants. MRT was only used with normal hearing individuals since the bilateral hearing-impaired and asymmetrical hearing-impaired participants had hearing thresholds over 25 dB HL, and therefore, would likely have struggled significantly to perform well on the test. Then, we would not have known if it was due to a weakness in the electrical signal or the participant's hearing loss causing the poor scores
Measure: Mean (Standard Deviation); unit: percentage of correct scores on MRT
Arm/Group | Normal Hearing Subjects | Bilateral Hearing Impaired | Asymmetrical Hearing-impaired
Number analyzed (Participants) | 20 | 0 | 0
percentage of correct scores on MRT
  Forehead | 84.38 (14.9) |  |
  Mastoid | 94.06 (5.9) |  |
  Neck | 84.06 (11.6) |  |

3. Primary Outcome: Speech Intelligibility in Quiet and Noisy Environments
Description: Measured using the modified rhyme test (MRT) consisting of a set of 50 six-item wordlist. Each word list contains single syllable words with a consonant-vowel-consonant sound sequence. Subjects completed electrical word recognition testing in a quiet, then a noisy environment. Electrodes were placed at 3 unique locations (mastoid, wrist, back) to measure how well speech could be delivered to the subject through the skin electrodes in a manner that would allow subjects to recognize words in a quiet and noisy environment. There were 2 experiments done for speech intelligibility. The first involved 20 subjects (outcome2) and aimed to assess speech intelligibility performance in a basic, quiet environment without background noise. This phase focused on evaluating the fundamental hearing performance. Once it was established that speech intelligibility was satisfactory with electrical stimulation, we proceeded to test an additional 30 subjects in both quiet and noisy environments (outcome3)
Time Frame: Baseline; approximately 2 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of correct MRT scores
Arm/Group | Normal Hearing Subjects | Bilateral Hearing Impaired | Asymmetrical Hearing-impaired
Number analyzed (Participants) | 30 | 0 | 0
percentage of correct MRT scores
  Mastoid-Quiet Environment | 93.86 (8.2) |  |
  Wrist-Quiet Environment | 93 (9.7) |  |
  Back-Quiet Environment | 93.83 (10.2) |  |
  Mastoid-Noisy Environment | 85.37 (11.7) |  |
  Wrist-Noisy Environment | 86 (12.7) |  |
  Back-Noisy Environment | 82.07 (12.5) |  |

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through study completion, approximately 2 hours.
Arm/Group | Normal Hearing Subjects | Bilateral Hearing Impaired | Asymmetrical Hearing-impaired
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/5 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/5 | 0/8
Other Adverse Events (participants affected / at risk) | 0/55 | 0/5 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2024-09-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT05112809/Prot_000.pdf